CLINICAL TRIAL: NCT05729295
Title: Cerebral Vascular Malformations: From Multimodal Imaging, to Endovascular, Surgical or Combined Treatment.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Alexandre Andrea, MD MSc, MD, MSc, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3957
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: AVM (Arteriovenous Malformation) Intracranial
MeSH Terms: conditions — Intracranial Arteriovenous Malformations | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endovascular embolization or surgery — Endovascular embolization with embolizing agents (including glue, non-adhesive agents) or neurosurgical excision of the lesion.

SUMMARY:
Cerebrovascular malformations (CVMs) are a heterogeneous group of disorders and can be classified histopathologically into five main categories: arteriovenous malformations (AVMs), dural arteriovenous fistulas (AVDs), abnormalities of venous development or venous angiomas (VAS), cavernous malformations (CVMs), ) and capillary telangiectasis (TAC). A further classification, more useful from a therapeutic point of view, is the functional one, which provides for a subdivision into two categories: CVD with arteriovenous shunt - among which AVMs and AVD stand out - and CVD without arteriovenous shunt.

AVMs and AVDs represent the two cerebrovascular malformations of greatest interest in the field of interventional neuroradiology. AVMs generally have a congenital origin, an estimated prevalence in the population of 0.005-0.6% and are most commonly diagnosed between the ages of 20 and 40, with an estimated annual bleeding risk between 4% and 4%; AVDs are rarer and have a predominantly acquired origin, in relation to previous thrombosis and trauma.

Intra- and extra-parenchymal hemorrhages are a frequent finding of cerebral vascular malformations, associated or not with headache, epileptic seizures or focal neurological deficits (from mass effect or vascular steal, with consequent ischemia); in this particular situation, the patient is subjected in the shortest possible time to a clinical-anamnestic assessment, to evaluate the severity of the clinical picture, which is followed by a tomographic examination to evaluate the extent of the lesions and classify the malformation- classification of Spetzler-Martin for AVMs and Cognard or Borden classification for AVDs.

Therefore, it is the authors' intention to conduct a retrospective and prospective observational study with the aim of exploring the possible implication of new variables that can predict with sufficient accuracy the outcome of patients with ruptured and unruptured cerebral vascular malformations; a possible positive response could be followed by a more structured clinical trial with which to derive the appropriate conclusions with greater methodological soundness.

DETAILED DESCRIPTION:
Cerebrovascular malformations (CVMs) are a heterogeneous group of disorders and can be classified histopathologically into five main categories: arteriovenous malformations (AVMs), dural arteriovenous fistulas (AVDs), abnormalities of venous development or venous angiomas (VAS), cavernous malformations (CVMs), ) and capillary telangiectasis (TAC). A further classification, more useful from a therapeutic point of view, is the functional one, which provides for a subdivision into two categories: CVD with arteriovenous shunt - among which AVMs and AVD stand out - and CVD without arteriovenous shunt.

AVMs and AVDs represent the two cerebrovascular malformations of greatest interest in the field of interventional neuroradiology. AVMs generally have a congenital origin, an estimated prevalence in the population of 0.005-0.6% and are most commonly diagnosed between the ages of 20 and 40, with an estimated annual bleeding risk between 4% and 4%; AVDs are rarer and have a predominantly acquired origin, in relation to previous thrombosis and trauma.

Intra- and extra-parenchymal hemorrhages are a frequent finding of cerebral vascular malformations, associated or not with headache, epileptic seizures or focal neurological deficits (from mass effect or vascular steal, with consequent ischemia); in this particular situation, the patient is subjected in the shortest possible time to a clinical-anamnestic assessment, to evaluate the severity of the clinical picture, which is followed by a tomographic examination to evaluate the extent of the lesions and classify the malformation- classification of Spetzler-Martin for AVMs and Cognard or Borden classification for AVDs.

Intra- and extra-parenchymal hemorrhages are a frequent finding of cerebral vascular malformations, associated or not with headache, epileptic seizures or focal neurological deficits (from mass effect or vascular steal, with consequent ischemia); in this particular situation, the patient is subjected in the shortest possible time to a clinical-anamnestic assessment, to evaluate the severity of the clinical picture, which is followed by a tomographic examination to evaluate the extent of the lesions and classify the malformation- classification of Spetzler-Martin for AVMs and Cognard or Borden classification for AVDs.

Numerous developments have been observed in the treatment, elective or acute, of AVMs and AVDs, ranging from neurosurgical intervention, endovascular embolization procedures using coils and adhesive and non-adhesive embolizing materials - even partial in view of a subsequent surgery - reaching to radiosurgical treatment (gamma-knife, cyber-knife and linear accelerator). Regardless of the type, the primary goal of treatment is healing, which occurs when the cerebral vascular malformation is permanently and persistently excluded from circulation.

Although clinical trials and meta-analyses have dispelled any doubts about the validity/necessity of the therapies, the authors are convinced that there may be some clinical and radiological characteristics, not fully explored in the aforementioned studies, which can help predict the outcome of such patients. The finding of these variables, if confirmed by subsequent trials aimed at the purpose, could in the future guide the selection of patients to undergo treatment as well as guide the choice of the best technique, endovascular or surgical in primis, to be applied according to the characteristics of each patient .

Therefore, it is the authors' intention to conduct a retrospective and prospective observational study with the aim of exploring the possible implication of new variables that can predict with sufficient accuracy the outcome of patients with ruptured and unruptured cerebral vascular malformations; a possible positive response could be followed by a more structured clinical trial with which to derive the appropriate conclusions with greater methodological soundness.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* unruptured and ruptured cerebral vascular malformation with consistent neurologic and radiologic evidence.
* Performing CT without contrast medium and CT angiography.
* Execution of an endovascular embolization procedure (which is indicated by a neurosurgeon and interventional neuroradiologist) or surgical treatment.

Exclusion Criteria:

- causes of haemorrhage other than cerebral vascular malformations (example: aneurysms and trauma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Given the purely descriptive nature of the primary objective, we do not proceed with the formal calculation of the sample size but a sample of N=200 patients is proposed.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Independence | 90 days clinical evaluation
  Functional independence at 90 days assessed by modified Rankin scale (mRS). A good clinical outcome will be defined as an mRS score between 0 and 2 (as per the literature).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A.Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexandre AM, Sturiale CL, Bartolo A, Romi A, Scerrati A, Flacco ME, D'Argento F, Scarcia L, Garignano G, Valente I, Lozupone E, Pedicelli A. Endovascular Treatment of Cavernous Sinus Dural Arteriovenous Fistulas. Institutional Series, Systematic Review and Meta-Analysis. Clin Neuroradiol. 2022 Sep;32(3):761-771. doi: 10.1007/s00062-021-01107-0. Epub 2021 Dec 15. PMID 34910224